CLINICAL TRIAL: NCT02108990
Title: Acetaminophen and Social Pain in Borderline Personality Disorder
Brief Title: Acetaminophen and Social Processes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Principal Investigator, Baldwin Way, Assistant Professor, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2012HO294; KL2RR025754-04 (NIH)
Record Dates: First submitted 2014-04-07; First posted 2014-04-09 (Estimated); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Borderline Personality Disorder
Keywords: borderline personality disorder; rejection; social pain
MeSH Terms: conditions — Borderline Personality Disorder; Rejection, Psychology | interventions — Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Acetaminophen 1000mg (Experimental): Acetaminophen 1000mg capsule orally three times a day
  Interventions: Drug: Acetaminophen

INTERVENTIONS:
Drug: Acetaminophen
  Other Names: Tylenol

SUMMARY:
Recent research has identified heightened sensitivity to social rejection as a core feature of BPD. Rejection sensitivity can trigger the aggressive, impulsive, and self-injurious behaviors characteristic of the disorder.

Therefore targeting therapy towards the reduction of rejection sensitivity may improve the low rates of effectiveness of current pharmacological and behavioral therapies. Therefore, this proposal tests a theoretically-based pharmacological approach that specifically targets the heightened sensitivity to rejection experienced by BPD patients.

In prior research with normal controls, it was shown that chronic treatment with the physical pain-killer acetaminophen (e.g. Tylenol) reduced both neural responses to social rejection (using fMRI) as well as self-reported feelings of rejection in a daily diary study.

It is the aim of this research project to determine if the over-the-counter analgesic, acetaminophen (active ingredient in Tylenol), can reduce symptoms and behaviors in BPD patients. The goal of this proposal is to use an open-label design to determine if acetaminophen improves symptoms in BPD patients.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of borderline personality disorder
* 18 years or older
* if on psychiatric medication, must be on a stable dose
* able to swallow tablets

Exclusion Criteria:

* current, primary substance abuse, particularly alcoholism
* current eating disorder
* history or current psychotic disorder
* suicidal ideation or behavior requiring imminent inpatient treatment
* pregnancy
* Participants whose medication has not been stable for more than 4 weeks
* Impaired liver function (> 1.25x the upper limit of the reference range)
* Conditions that can affect immune system functioning.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2013-09; Primary Completion 2014-06-30 (Actual); Study Completion 2014-06-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in symptom reports on the PAI-BOR at week 6 | Baseline, Week 6
  Symptom reports on the PAI-BOR.
Change from baseline in symptom severity on the Zanarini Rating Scale for Borderline Personality Disorder | Baseline, Week 6
  Zanarini Rating Scale for Borderline Personality Disorder

SECONDARY OUTCOMES:
Symptom Reports | Baseline, weeks, 1,2,3,4,5,6 and 8.
  Each week participants will be emailed a link to complete that will have three surveys.
  1. The Beck Depression Inventory
  2. The Beck Anxiety Inventory
  3. The Inventory of Interpersonal Problems (Aggression and Interpersonal Sensitivity Subscales).
  This weekly survey report will also be sent to the participants once after the completion of pharmacotherapy (at the two weeks post cessation treatment).
Daily Diary | Daily for week 0,1,2, and 3
  The importance of these measures will be to assess how rejected, aggressive, and social participants have been in order to determine if acetaminophen affects these proclivities. Participants will report on: hurt feelings, rejection, affect, aggressive feelings, impulsive behaviors, alcohol use, sleep, social interactions, perceived stress, self-esteem

CONTACTS AND LOCATIONS:
Overall Officials: Baldwin M Way, Ph.D., Principal Investigator — Ohio State University; Jennifer S. Cheavens, Ph.D., Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

REFERENCES:
- [Background] Dewall CN, Macdonald G, Webster GD, Masten CL, Baumeister RF, Powell C, Combs D, Schurtz DR, Stillman TF, Tice DM, Eisenberger NI. Acetaminophen reduces social pain: behavioral and neural evidence. Psychol Sci. 2010 Jul;21(7):931-7. doi: 10.1177/0956797610374741. Epub 2010 Jun 14. PMID 20548058